CLINICAL TRIAL: NCT05269563
Title: Double Flap Technique Utilizing ERM and ILM for Macular Hole
Brief Title: Double Flap Technique for Macular Hole
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Omer Othman Abdullah (Other)
Responsible Party: Sponsor-Investigator, Omer Othman Abdullah, Associate consultant ophthalmologist, Ibinsina Modern Eye and Retina Center
Organization: Ibinsina Modern Eye and Retina Center (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IMER 11
Record Dates: First submitted 2022-01-28; First posted 2022-03-08 (Actual); Last update posted 2023-03-24 (Actual); Status verified 2023-03

CONDITIONS: Macular Holes
Keywords: Double Flaps
MeSH Terms: conditions — Retinal Perforations | interventions — Surgical Procedures, Operative

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Double flap technique to secure macular hole closure. (Experimental): Single ILM flap technique is already performing worldwide; however, sometimes it is associated with flap displacement. To overcome this issue, the double flap technique was tried.
  Interventions: Other: Surgical intervention

INTERVENTIONS:
Other: Surgical intervention — Pars Plana Vitrectomy for Macular Hole Closure

SUMMARY:
Double flapping technique to close the macular hole.

DETAILED DESCRIPTION:
Recently, it is agreed to close the macular hole with the retinal innermost layer; which is called internal limiting membrane (ILM), in most cases, the hole closes. But, sometimes the ILM single flap might displace resulting in a persistent hole.

Therefore, the investigators tried to make two flaps utilizing ILM, and sometimes certain patients have a very thin membrane over the retina; it is called epiretinal membrane (ERM). The investigators use the double flapping technique by utilizing ERM; therefore, the ILM remains and can be used if the hole resists closing with the first surgical interventions.

Here, the investigators did not use any new materials with unknown side effects on the human retina. Although the flap technique is well known; however, investigators are making a double flap to decrease the chance of persisting macular holes.

The visual recovery will be appeared in the post-operative period, whether it is the same, better, or worse.

ELIGIBILITY:
Inclusion Criteria:

* Full thickness macular hole

Exclusion Criteria:

* Partial-thickness macular hole
* Vitreomacular traction

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2023-03-23 (Actual); Study Completion 2023-03-23 (Actual)

PRIMARY OUTCOMES:
Ocular coherence tomography | The fourth week post-operatively
  The closure of the hole can be assessed clearly

CONTACTS AND LOCATIONS:
Overall Officials: Omer Abdullah, M.Sc., Principal Investigator — Ibinsina Modern Eye and Retina Center
Locations (1):
- Ibinsina Modern eye and retina center, Erbil, Iraq